CLINICAL TRIAL: NCT06413758
Title: Effect of Internal and External Focus on Balance Performance: Comparison of Virtual Reality and Real World Environment
Brief Title: Attentional Focus in Virtual Reality
Status: Not yet recruiting | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Aybike Senel, Research assistant, PT, PhD(c), Istanbul University - Cerrahpasa
Other Study IDs: 06052024
Record Dates: First submitted 2024-05-09; First posted 2024-05-14 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Attentional Focus in Virtual Reality
Keywords: Postural Control; Virtual Reality; Focus of Attention

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group I-Virtual Reality: In this group, participants will be in a virtual environment with a VR glass put on. The balance performance of the participants will be assessed with single leg stance test and bipodal stance test. The participants will be instructed to stand still and maintain balance on the forceplate in three conditions: (1) with an internal focus, (2) with an external focus, and (3) non-directional. Conditions will be applied to the participants randomly to avoid bias. Each condition will be measured three times and the mean values will be recorded as outcomes. The total displacement of center of pressure (CoP), the mean velocity of CoP, the CoP area, total mediolateral (ML) displacement, the mean velocity in ML, total anteroposterior (AP) displacement and the mean velocity in AP will assessed with K-Force Plates (Kinvent, France).
- Group II-Real World: The balance performance of the participants will be assessed with single leg stance test and bipodal stance test. The participants will be instructed to stand still and maintain balance on the forceplate in three conditions: (1) with an internal focus, (2) with an external focus, and (3) non-directional. Conditions will be applied to the participants randomly to avoid bias. Each condition will be measured three times and the mean values will be recorded as outcomes. The total displacement of center of pressure (CoP), the mean velocity of CoP, the CoP area, total mediolateral (ML) displacement, the mean velocity in ML, total anteroposterior (AP) displacement and the mean velocity in AP will assessed with K-Force Plates (Kinvent, France).

SUMMARY:
The goal of this explorative observational study is to learn about the effect of internal and external focus on postural control in virtual reality and compare with the real world environment in young adults. The main question it aims to answer is:

Does attentional focus effect differently on postural control in virtual reality comparing to real world environment?

DETAILED DESCRIPTION:
Virtual Reality is used to improve postural control in various populations. However, exercise with virtual reality glasses cause new challenges to the user in maintaining balance. In this study, the effect of internal and external focus on postural control in the virtual reality environment will be revealed and compared with the performance in the real environment. The results of the study will guide the customization and optimization of balance training programs implemented in the virtual reality environment. A total of 38 healthy young adults will be included and allocated into Group I (Virtual Reality) or Group II (Real World) (ratio 1:1). The balance performance of the participants will be assessed with single leg stance test and bipodal stance test. The participants will be instructed to stand still and maintain balance on the forceplate in three conditions: (1) with an internal focus, (2) with an external focus, and (3) non-directional. Conditions will be applied to the participants randomly to avoid bias. Each condition will be measured three times and the mean values will be recorded as outcomes. The total displacement of center of pressure (CoP), the mean velocity of CoP, the CoP area, total mediolateral (ML) displacement, the mean velocity in ML, total anteroposterior (AP) displacement and the mean velocity in AP will assessed with K-Force Plates (Kinvent, France).

ELIGIBILITY:
Inclusion Criteria:

* Being a healthy individual between the ages of 18-26
* Lower extremity functional motor signs or sensory features should be normal or corrected
* No lower extremity injury within 6 months
* Not taking alcohol or medication 12 hours before
* Having no virtual reality experience

Exclusion Criteria:

* History of epilepsy, marked dissociative seizures
* Needing assistive devices to maintain upright posture
* Other comorbidities that may affect postural control (dizziness, vestibular disorders, orthopedic or cardiovascular comorbidities)
* Being an athlete
* Positive Fukuda stepping test

Ages: 18 Years to 26 Years | Sex: All
Age Groups: Adult
Study Population: healthy young adults between the ages of 18-26
Sampling Method: Probability Sample
Enrollment: 38 (Estimated)
Dates: Start 2024-11-30 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-01-15 (Estimated)

PRIMARY OUTCOMES:
Total displacement of center of pressure | baseline
  Total displacement of center of pressure on the force plate
The mean velocity of center of pressure | baseline
  the mean velocity of center of pressure on the force plate
The area of center of pressure | baseline
  the area drawn by the movement of center of pressure on the force plate
total mediolateral displacement | baseline
  total mediolateral displacement of center of pressure on the force plate
total anterolateral displacement | baseline
  total anterolateral displacement of center of pressure on the force plate
the mean velocity in mediolateral | baseline
  the mean velocity of total mediolateral displacement of center of pressure on the force plate
the mean velocity in anterolateral | baseline
  the mean velocity of total anterolateral displacement of center of pressure on the force plate